CLINICAL TRIAL: NCT03046394
Title: Comparison Between Three Types of Prosthetic Feet: a Randomized Double-blind Controlled Single-subject Multiple-rater Trial
Brief Title: Comparison Between Three Types of Prosthetic Feet
Acronym: ProSto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: URIS201701
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Amputation; Traumatic, Leg, Lower, Between Knee and Ankle
Keywords: prosthetic feet; gait pattern; one leg standing; walking speed

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- C-SACH (Active Comparator): All the interventions will be administered to the patient in this single-subject trial, each 6 times
  Interventions: Device: C-SACH
- B-DER (Active Comparator): All the interventions will be administered to the patient in this single-subject trial, each 6 times
  Interventions: Device: B-DER
- A-DER (Active Comparator): All the interventions will be administered to the patient in this single-subject trial, each 6 times
  Interventions: Device: A-DER

INTERVENTIONS:
Device: C-SACH — Solid Ankle Cushion Heel by Otto Bock, advertised for activity category 1
  Arms: C-SACH
Device: B-DER — Dynamic Motion by Otto Bock, advertised for activity category 2-3
  Arms: B-DER
Device: A-DER — Triton by Otto Bock, advertised for activity category 3-4
  Arms: A-DER

SUMMARY:
One Solid Ankle Cushion Heel (SACH) and two Dynamic Elastic Response (DER) prosthetic feet will be tried six times in random order by the patient. The patient will be an active prosthetic foot user who walks several kilometers per day and was amputated at the trans-tibial level because of injury. Gait pattern will be rated in comparison with the patient's previous prosthetic foot by a physiatrist, physiotherapist, prosthetist and the patient. One-leg standing and 10-meter walking tests will also be performed.

DETAILED DESCRIPTION:
The prosthetic feet will be: one SACH foot (by Otto Bock - foot C, advertised for activity category 1) and two DER feet (Dynamic Motion by Otto Bock - foot B, advertised for activity category 2-3; and Triton by Otto Bock - foot A, advertised for activity category 3-4).

All the prosthetic feet are of the same size and chosen for the patient's weight. They will be covered so that neither the patient nor professionals will be able to see which prosthetic foot is being used.

The study is blinded because the prosthetist designated for changing the prosthetic feet will be the only one who will know which prosthetic is being used. The orientational sample size calculation and the randomisation plan were prepared by a statistician.

The first trial will be performed using the patient's own prosthetic foot in order to establish a baseline. The patient will then have to to compare the prosthetic feet with his own existing prosthetic foot and rate the ability to walk on even terrain (100m), uneven terrain (grass, 100m), decline and incline (i.e., slope), and up and down the stairs (one floor) on a five-point Likert-type scale (-2 much worse, -1 slightly worse, 0 the same, 1 slightly better, 2 much better). After each trial he will also perform the one-leg standing test (with three repetitions) and the 10-meter walking test. Before each trial, the patient will be given 15 minutes for adaptation to each new prosthetic foot without the presence of the assessors.

The three expert observers will be: a physical and rehabilitation medicine specialist physician, a certified prosthetist-orthotist, and a physiotherapist. Each has got over 20 years of experience in rehabilitation of patients after amputation and observation of their gait. They will be blind to the currently used prosthetic foot. They will follow the patient and assess his walking using the same rating scale in comparison with the initial trial as the patient.

ELIGIBILITY:
Inclusion Criteria:

* active prosthetic foot user who walks several kilometers per day
* amputation at the trans-tibial level >5 years ago

Exclusion Criteria:

* other medical problems

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Rating | Immediately after each trial
  Likert-type, compared to the patient's existing prosthetic foot (-2 much worse, -1 slightly worse, 0 the same, 1 slightly better, 2 much better)

SECONDARY OUTCOMES:
The time that the patient can stand on the prosthetic foot | Immediately after the rating, repeated 3 times
  Measured by the one-leg standing test (average of three repetitions)
Walking velocity | Immediately after the one-leg standing test
  Measured by the 10-meter walking test

CONTACTS AND LOCATIONS:
Overall Officials: Helena Burger, MD, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No